CLINICAL TRIAL: NCT05090202
Title: Prevalence of Prediabetes and Newly Diagnosed Diabetes in Patients With HFpEF( Heart Failure With Preserved Ejection Fraction) and HFrEF(Heart Failure With Reduced Ejection Fraction) in Sohag University Hospital
Brief Title: Prediabetes and Newly Diagnosed Diabetes in Chronic Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Heba Saber AbdelKader, Principal Investigator, Sohag University
Other Study IDs: diabetes and heart failure
Record Dates: First submitted 2021-09-13; First posted 2021-10-22 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HFrEF " Heart failure with reduced ejection fraction": chronic heart failure with echocardiographic finding of LVEF "Left ventricular ejection fraction" equal or less than 40%
  Interventions: Diagnostic Test: hbA1C
- HFmrEF "Heart failure with mildly reduced ejection fraction": chronic heart failure with echocardiographic finding of LVEF between 41% and 49%
  Interventions: Diagnostic Test: hbA1C
- HFpEF " Heart failure with preserved ejection fraction": chronic heart failure with echocardiographic finding of LVEF equal or more than 50%
  Interventions: Diagnostic Test: hbA1C

INTERVENTIONS:
Diagnostic Test: hbA1C — hbA1C will be measured for all patients and results will be analysed into Non diabetic, Prediabetic and Diabetic

SUMMARY:
The aim the study is to determine the prevalence of prediabetic dysglycemia and newly diagnosed diabetes among individuals with CHF(chronic heart failure) in sohag university hospital patients .

DETAILED DESCRIPTION:
- Prospective study to:

1. study the differences in the prevalence of Prediabetes and newly diagnosed diabetes among the patients with HFrEF and HFpEF
2. The effect of dysglycemia on prognosis of patients with chronic heart failure.
3. The effect of early discover of diabetes mellitus on prognosis of patients with chronic heart failure

ELIGIBILITY:
Inclusion criteria:

* All patients presented by heart failure
* 18 years or older
* Classified according to NYHA " New York Heart Association" classification from NYHA class 2 and more

Exclusion Criteria:

* Overt diabetes
* Rheumatic Heart Disease
* Congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presented by heart failure NYHA class 2 or more and admitted to Sohag University hospital according to inclusion and exclusion criterea
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Heart failure hospitalization. | From date of randomization up to 1 month
  Heart failure hospitalization or cardiovascular (CV) death, and all-cause death, and estimated hazard ratios (HR) by use of multivariable Cox regression models.

REFERENCES:
- [Background] Nielsen R, Jorsal A, Iversen P, Tolbod L, Bouchelouche K, Sorensen J, Harms HJ, Flyvbjerg A, Botker HE, Wiggers H. Heart failure patients with prediabetes and newly diagnosed diabetes display abnormalities in myocardial metabolism. J Nucl Cardiol. 2018 Feb;25(1):169-176. doi: 10.1007/s12350-016-0622-0. Epub 2016 Jul 29. PMID 27473218